CLINICAL TRIAL: NCT00600405
Title: The Efficacy of Tamsulosin in the Treatment of Ureteral Stones in Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Maine Medical Center Mentored Research Committee (Unknown)
Responsible Party: Andrew Perron, MD, Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2958
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Nephrolithiasis; Ureteral Calculi
Keywords: Nephrolithiasis; Ureteral Calculi
MeSH Terms: conditions — Nephrolithiasis; Ureteral Calculi | interventions — Tamsulosin; Standard of Care; Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Subjects randomized to the experimental group receive ibuprofen, oxycodone, and tamsulosin 0.4 mg orally daily for ten days.
  Interventions: Drug: tamsulosin
- II (Other): Standard therapy arm: subjects randomized to standard therapy receive ibuprofen and oxycodone alone.
  Interventions: Drug: Standard therapy with ibuprofen and oxycodone.

INTERVENTIONS:
Drug: tamsulosin — Tamsulosin 0.4 mg orally daily for ten days.
  Other Names: Flomax
  Arms: I
Drug: Standard therapy with ibuprofen and oxycodone. — Oxycodone: 5mg, one to two tablets every four to six hours as needed for pain. Ibuprofen: 800 mg, one three times a day with food as needed for pain.
  Arms: II

SUMMARY:
The purpose of this study is to determine the efficacy of the α-adrenergic antagonist tamsulosin in the treatment of adult emergency department (ED) patients with ureteral colic secondary to lower ureteral calculus. We hypothesize that there will be no difference in outcomes for subjects treated with and without tamsulosin.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial seeks to compare outcomes for adult emergency department patients with lower ureteral calculus. Subjects will be randomized to receive treatment with ibuprofen and oxycodone alone (standard therapy) or standard therapy plus tamsulosin 0.4mg orally once daily for ten days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* able to read, write, and speak English;
* able to use the NRS pain scale; and
* computed tomography diagnosed single lower ureteral calculus

Exclusion Criteria:

* allergy or sensitivity to the study drug (tamsulosin hydrochloride [Flomax]);
* sulfa/sulfonamide allergy;
* inability to provide informed consent;
* lithiasis of the ureteral intramural tract;
* acute or chronic renal failure;
* fever;
* presence of multiple ureteral stones;
* peptic ulcer disease;
* liver failure;
* concomitant treatment with alpha-lytic drugs, calcium antagonists, nitrates, or vardenafil (Levitra);
* pregnancy;
* breastfeeding; or
* a history of urinary surgery or endoscopic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Rate of spontaneous ureteral stone expulsion | 48, 120, 336 hours

SECONDARY OUTCOMES:
Time to spontaneous ureteral stone expulsion. | 48, 120, 336 hours
Self-reported NRS-11 pain scores. | 48, 120, 336 hours
Number of colicky pain episodes. | 48, 120, 336 hours
Number of days missed work or usual functional ability. | 48, 120, 336 hours
Number of return ED visits or unscheduled PCP visits for continued pain. | 48, 120, 336 hours
Amount of narcotic pain medication used. | 48, 120, 336 hours
Adverse medication-related events. | 48, 120, 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Perron, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States